CLINICAL TRIAL: NCT05502627
Title: To Study the Healing Effect of 0.25% Lemongrass Oil Mouthwash on Chronic Periodontitis Patients by Evaluating the Levels of Transforming Growth Factor-beta
Brief Title: To Study the Healing Effect of 0.25% Lemongrass Oil Mouthwash on Chronic Periodontitis Patients.
Status: Completed | Type: Observational
Sponsor: Postgraduate Medical Institute, Lahore (Other)
Responsible Party: Principal Investigator, Ummara Komal, Doctor, Postgraduate Medical Institute, Lahore
Other Study IDs: PGMILahorePakistan
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: scaling was done along with intervention (0.25% lemongrass mouthwash was given)
  Interventions: Drug: 0.25% lemon grass oil mouthwash
- control group: only scaling was done

INTERVENTIONS:
Drug: 0.25% lemon grass oil mouthwash — 0.25% lemon grass oil mouth wash given twice daily for fourteen days to the patients of chronic periodontitis after scaling in experimental group and in control group only scaling was done.
  Other Names: lemon grass mouth wash
  Groups: Experimental group

SUMMARY:
Periodontitis is the inflammation of the tissues supporting the teeth. Lemongrass (Cymbopogon Citratus) oil mouthwash can be used with subgingival scaling in the treatment of periodontal diseases. Transforming growth factor beta (TGF-β) is a multifunctional cytokine belonging to transforming growth factor superfamily and its elevated levels are detectable in inflammatory and healing process The present project will be conducted to evaluate the expression of TGF-β levels in chronic periodontitis patients after ultrasonic scaling and using 0.25% lemongrass oil mouthwash. TGF-β is a salivary marker of periodontitis.

DETAILED DESCRIPTION:
Periodontitis is the inflammation of the tissues supporting the teeth which include cementum, gingiva, periodontal ligaments and alveolar bone. Periodontitis typically follows untreated gingivitis, a shift in the composition of biofilm from gram positive cocci to dominantly gram negative actinomyces and infection by proteolytic obligate anaerobes resulting in progressive destruction of periodontal ligament, formation of pocket around the teeth and resorption of alveolar bone with ultimately loosening or loss of teeth. The present project will be associated with very common forms of periodontitis (in which the inflammation results in periodontal tissue destruction and alveolar bone resorption) and gingivitis (in which the inflammation is confined to gingivae and is reversible with good oral hygiene). Lemongrass (Cymbopogon Citratus) oil mouthwash can be used with subgingival scaling to eliminate the pathogens of periodontitis and to treat the inflammation and the damage done to periodontium by it. It possess anti-oxidant, anti-inflammatory, anti-microbial, anti-fungal and astringent properties. Citral epoxide which is an ingredient of lemongrass extract is an active anti-inflammatory and anti-bacterial agent. It is useful in dentistry and has a wide role in the treatment of periodontal diseases. Transforming growth factor beta (TGF-β) is a multifunctional cytokine belonging to transforming growth factor superfamily and its elevated levels are detectable in inflammatory and healing process The present project will be conducted to evaluate the expression of TGF-β levels in chronic periodontitis patients after ultrasonic scaling and using 0.25% lemongrass oil mouthwash. TGF-β is a salivary marker of periodontitis. A sample size of 30 patients either male or female aged between 40 and 60 years with chronic localized or generalized periodontitis with pocket depth of >3mm affecting at least two nonadjacent sites/teeth will be selected. This sample will be divided into two equal groups. In the experimental 1 group, only sub-gingival scaling will be performed. In the experimental 2 group, sub-gingival scaling will be performed, followed by use of 0.25% lemongrass oil mouthwash twice daily for 14 days. Saliva sample will be collected on days 0, 7 and 14 and level of salivary biomarker, TGF-β will be measured with the ELISA technique. The data will be entered and analyzed using SPSS 22. Mean ±SD will be given for quantitative variables like TGF-β level. A p value of ≤ 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age between 40-60 years with generalized periodontitis
2. Minimum 15 teeth should present in oral cavity
3. Patient who don't have received periodontal therapy for last three months
4. Probing depth > 3mm

Exclusion Criteria:

1. Patient taking antibiotics or NSAIDS within last three months
2. Patients with oral mucous lesions, Oral carcinoma, xerostomia, previous history of radiotherapy or chemotherapy
3. Hypersensitivity to lemongrass
4. Any systemic illness
5. Pregnant females

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female with age range between 40-60 years with generalized periodontitis were taken for the study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
To observe the healing of patients with chronic periodontitis. | 10 months
  0.25% lemon grass oil effect on healing of chronic periodontitis by measuring levels of TGF-Beta.

CONTACTS AND LOCATIONS:
Overall Officials: Asrar Ahmed, M. Phil. OB, Study Director — PGMI, Lahore
Locations (1):
- Punjab dental hospital, Lahore, Punjab Province, Pakistan